CLINICAL TRIAL: NCT00813488
Title: A Double Blind, Active Controlled Crossover Study to Evaluate the Efficacy and Safety of Fentanyl Buccal Tablets Versus Immediate Release Oxycodone for the Management of Breakthrough Pain in Opioid Tolerant Patients With Chronic Pain
Brief Title: Fentanyl Buccal Tablets Versus Immediate Release Oxycodone for Breakthrough Pain in Patients With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C25608/3056/BP/US
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Results first posted 2010-12-31 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Pain
Keywords: Breakthrough Pain; Opioid-tolerant; Chronic Pain
MeSH Terms: conditions — Chronic Pain; Breakthrough Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fentanyl buccal tablet first then immediate release oxycodone (Experimental): This crossover study includes a screening period, two titration periods, two double-blind treatment periods during which subjects will be randomized to receive fentanyl buccal tablet (FBT) plus placebo during the first treatment period and then immediate release oxycodone plus placebo during the second treatment period or vice versa, then followed by a 12-week open-label treatment period with FBT or an alternative short acting opioid.
  Interventions: Drug: Fentanyl Buccal Tablet; Drug: Immediate release oxycodone
- Immediate Release Oxycodone first then FBT (Experimental): This crossover study includes a screening period, two titration periods, two double-blind treatment periods during which subjects will be randomized to receive fentanyl buccal tablet (FBT) plus placebo during the first treatment period and then immediate release oxycodone plus placebo during the second treatment period or vice versa, then followed by a 12-week open-label treatment period with FBT or an alternative short acting opioid.
  Interventions: Drug: Fentanyl Buccal Tablet; Drug: Immediate release oxycodone

INTERVENTIONS:
Drug: Fentanyl Buccal Tablet — FBT dose strengths = 200, 400, 600, or 800 mcg (1, 2, 3, or 4 tablets) taken prn (as needed) in the event of breakthrough pain.
  The maximum dose of FBT permitted during the titration and double-blind periods in this study is 800 mcg (4 tablets).
  For the subsequent 12-week open-label treatment period, patients will either continue with FBT treatment or begin treatment with an alternative short-acting opioid deemed appropriate for each patient by the clinician.
  Other Names: CEP-25608
Drug: Immediate release oxycodone — Immediate release oxycodone dosage strength: 15, 30, 45, and 60 mg doses (1, 2, 3 or 4 capsules) to be taken prn (as needed) for breakthrough pain.
  The maximum single dose would be 60 mg (4 capsules).

SUMMARY:
Evaluate the efficacy of treatment with the fentanyl buccal tablet (FBT) compared with immediate release oxycodone treatment in alleviating breakthrough pain (BTP) in opioid tolerant patients with chronic pain.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has chronic pain of at least 3 months duration associated with any of the following conditions: diabetic peripheral neuropathy, postherpetic neuralgia, traumatic injury, complex regional pain syndrome, back pain, neck pain, fibromyalgia, chronic pancreatitis, osteoarthritis, rheumatoid arthritis, or cancer. Other chronic painful conditions may be evaluated for possible inclusion.
* The patient is currently using at least one of the following: at least 60 mg of oral morphine/day, or at least 25 mcg of transdermal fentanyl/hour, or at least 30 mg of oxycodone/day, or at least 8 mg of hydromorphone/day, or an equianalgesic dose of another opioid/day as ATC therapy for at least 7 days before administration of the first dose of study drug.
* The patient is willing to provide written informed consent, including a written opioid agreement form, to participate in this study.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of birth control and agree to continued use of this method for the duration of the study.
* Any patient with cancer should have a life expectancy of at least 3 months.
* The patient reports an average PI score, over the 24 hours prior to screening, of 6 or less (0=no pain through 10=pain as bad as you can imagine) for their chronic pain.
* The patient experiences, on average, at least 1 and less than 5 BTP episodes per day while taking ATC opioid therapy, and on average, the duration of each BTP episode is less than 4 hours during the screening period.
* The patient currently uses opioid therapy for alleviation of BTP episodes, occurring at the location of the chronic pain, and achieves at least partial relief.
* The patient must be willing and able to successfully self administer the study drug, comply with study restrictions, complete the electronic diary, and return to the clinic for scheduled study visits as specified in this protocol.

Key Exclusion Criteria:

* The patient has uncontrolled or rapidly escalating pain as determined by the investigator or has pain uncontrolled by therapy that could adversely impact the safety of the patient or that could be compromised by treatment with study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in either study drug.
* The patient has a diagnosis of chronic headache or migraine as the primary painful condition with associated BTP.
* The patient has cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with potent synthetic opioids.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise the patient's safety or collected data.
* The patient has suicidal ideation at screening or has a history of suicidal ideation within 1 year or history of suicide attempt within 2 years before screening, or a diagnosis of bipolar disorder or history of schizophrenia
* The patient is expected to have surgery during the study that will impact the patient's chronic pain and/or BTP.
* The patient has had therapy before study drug treatment that, in the opinion of the investigator, could alter pain or response to pain medication.
* The patient is pregnant or lactating.
* The patient has participated in a previous study with FBT.
* The patient has participated in a study involving an investigational drug in the prior 30 days.
* The patient is currently using FBT or oral transmucosal fentanyl citrate for BTP.
* The patient is currently using immediate-release oxycodone for BTP and is unwilling to undergo re-titration.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (e.g., regional nerve block) that could, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise collected data.
* The patient is involved in active litigation in regard to the chronic pain currently being treated.
* The patient has a positive UDS for an illicit drug or a medication not prescribed for him/her or which is not medically explainable (i.e., active metabolites).
* The investigator feels that the patient is not suitable for the study for any reason (e.g., the patient's social history indicates an increased risk of drug diversion)
* Additional exclusion criteria will apply for patients who decide to participate in the pharmacokinetics assessment to be performed at designated study sites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon
Locations (50):
- United States (50):
  - Parkway Medical Center, Birmingham, Alabama
  - Horizon Research Group, Inc, Mobile, Alabama
  - Robert Karns, MD a Medical Corporation, Beverly Hills, California
  - Catalina Research Institute, LLC, Chino, California
  - Pacific Coast Pain Management, Laguna Hills, California
  - Loma Linda University Health, Loma Linda, California
  - VA Northern California Health, Mather, California
  - New England Research Associates, Trumbull, Connecticut
  - Delray Research Associates, Delray Beach, Florida
  - Emerald Coast Research Group Inc, Marianna, Florida
  - Compass Research, LLC, Orlando, Florida
  - Gold Coast Research, Plantation, Florida
  - Sarasota Pain Medicine Research, Sarasota, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Taylor Research, Marietta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Georgia Pain Care, Newnan, Georgia
  - South Coast Medical Group, Savannah, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - Suburban Clinical Research, Bolingbrook, Illinois
  - Knight Center for Integrated Health, Peoria, Illinois
  - Indiana Medical Research, Elkhart, Indiana
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - Indiana Pain & Spine Clinic, South Bend, Indiana
  - ICRI Inc., Overland Park, Kansas
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Gulf Coast Research Associates, Inc, Baton Rouge, Louisiana
  - Columbia Medical Practice, Columbia, Maryland
  - MidAtlantic Pain Medicine Center, Pikesville, Maryland
  - Michigan Neurology Associates PC, Clinton Township, Michigan
  - CRC of Jackson, Jackson, Mississippi
  - Healthcare Research, Florissant, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Clinical Research Source Inc, Perrysburg, Ohio
  - Pain Research of Oregon, Eugene, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Research Center, West Reading, Pennsylvania
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Trident Institute of Medical Research, LLC, North Charleston, South Carolina
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Lovelace Scientific, Austin, Texas
  - Sun Research Institute, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah

REFERENCES:
- [Derived] Webster LR, Slevin KA, Narayana A, Earl CQ, Yang R. Fentanyl buccal tablet compared with immediate-release oxycodone for the management of breakthrough pain in opioid-tolerant patients with chronic cancer and noncancer pain: a randomized, double-blind, crossover study followed by a 12-week open-label phase to evaluate patient outcomes. Pain Med. 2013 Sep;14(9):1332-45. doi: 10.1111/pme.12184. Epub 2013 Jul 15. PMID 23855816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with chronic pain who had been receiving opioid therapy for the previous 7 days and reported on average 1 to 5 breakthrough pain episodes per day were recruited from 50 different study sites throughout the United States beginning December 2008 and completing in November 2009.
Pre-assignment Details: Prior to the double-blind treatment period, subjects participated in two titration periods to identify a "successful" and tolerated dose of FBT and immediate-release oxycodone. Subjects who did not titrate to a successful and tolerated dose were excluded from further participation in the study.
Groups:
- FBT First Immediate Release Oxycodone Second: Subjects in this treatment group were assigned 200 mcg FBT during the first titration period and then 15 mg oxycodone during the second titration period. Standard rescue medication could be taken if pain relief was unsuccessful. If more than one dose was required for at least 1 of 3 breakthrough pain episodes in one day, the next day the dose was increased (in 200 mcg increments for FBT and 15 mg increments for oxycodone). The maximum allowable dose was 800 mcg for FBT (4 tablets) and 60 mg (4 capsules) for oxycodone. If a dose was not tolerated the dose was lowered to the previous tolerated dose. Titration completed when successful analgesia was achieved with a tolerated dose or maximum dose was reached. If unsuccessful at maximum dose subject was discontinued from proceeding further in the study. Subjects who successfully titrated were randomized.
- Immediate-Release Oxycodone First FBT Second: Subjects in this treatment group were assigned 15 mg oxycodone during the first titration period and then 200 mcg FBT during the second titration period. Standard rescue medication could be taken if pain relief was unsuccessful. If more than one dose was required for at least 1 of 3 breakthrough pain episodes in one day, the next day the dose was increased (in 200 mcg increments for FBT and 15 mg increments for oxycodone). The maximum allowable dose was 800 mcg for FBT (4 tablets) and 60 mg (4 capsules) for oxycodone. If a dose was not tolerated the dose was lowered to the previous tolerated dose. Titration completed when successful analgesia was achieved with a tolerated dose or maximum dose was reached. If unsuccessful at maximum dose subject was discontinued from proceeding further in the study. Subjects who successfully titrated were randomized.
Period: Titration Period 1
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 107 | 106
Completed | 80 | 89
Not Completed | 27 | 17
Not completed — Adverse Event | 6 | 1
Not completed — Lack of Efficacy | 9 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 4 | 3
Not completed — Non-compliance to study medication | 4 | 1
Not completed — Non-compliance to study procedures | 2 | 2
Not completed — Technical Difficulties | 0 | 1
Period: Titration Period 2
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 80 | 89
Completed | 64 | 79
Not Completed | 16 | 10
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 8 | 4
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance with study procedures | 2 | 1
Period: Double-blind Treatment Period 1
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 72 (After titration subjects were re-randomized to these two treatment arms) | 71 (After titration subjects were re-randomized to these two treatment arms)
Completed | 71 | 66
Not Completed | 1 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: Double-blind Treatment Period 2
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 71 | 66
Completed | 66 | 65
Not Completed | 5 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Other | 1 | 0
Period: Open-label Extension
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 65 (Patients completing double-blind periods were randomized to FBT or standard of care for open-label) | 66 (Patients completing double-blind periods were randomized to FBT or standard of care for open-label)
Completed | 53 (This group received FBT open--label) | 59 (This group received standard of care (including immediate-release oxycodone))
Not Completed | 12 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Non-compliance study medication | 4 | 0
Not completed — Non-compliance study procedures | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Number of Patients
Number analyzed (Participants) | 213
Age Continuous [Mean (Standard Deviation); unit: years] | 51.0 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 195
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 191
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 213
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (7.25)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Difference (PID) at 15 Minutes Post-treatment (PID15)
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID15 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 15 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and 15 minutes after dosing
Population: Full Analysis Set defined as having at least one evaluable episode of breakthrough pain treated with FBT and at least one with oxycodone. An episode was evaluable if it had a valid pain intensity measurement immediately prior to drug administration. No imputation for missing breakthrough pain episodes, but LOCF was applied for missing PI scores.
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Units Other Than Participants: Breakthrough pain episodes
Groups:
- Fentanyl Buccal Tablet (FBT): FBT or matching placebo during the 2 double-blind treatment periods at doses of 200, 400, 600, and 800 mcg was self-administered by patients.
  PTs were initially titrated with FBT during the 1st titration period and immediate release oxycodone during the 2nd titration period or immediate-release oxycodone in the 1st titration period then FBT in the 2nd titration period.
  During the 12-week open-label extension period, pts randomized to FBT treatment were initially dispensed single tablets at the dose found to be successful during the titration period.
- Immediate-release Oxycodone (OXY): Immediate-release oxycodone (or matching placebo) at doses of 15,30, 45, and 60 mg was self administered. The double-blind, treatment period used a 2 period crossover design in which the patient first managed 10 episodes with 1 of the 2 blinded study drugs (successful doses of immediate-release oxycodone or FBT) and then managed a subsequent 10 episodes with the other blinded study drug.
  Patients were initially titrated to immediate-release oxycodone during the 1st titration period and to FBT during the 2nd titration period or to FBT during the 1st titration period and immediate-release oxycodone during the 2nd titration period.
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on scale | 0.88 (0.09) | 0.76 (0.09)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID15 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p = 0.0004, Mixed effects ANOVA crossover model; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.06 to 0.20], Standard Error of Mean 0.09

2. Secondary Outcome: Pain Intensity Difference (PID) at 5 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID5 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 5 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and 5 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | .08 (.02) | .06 (.02)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID5 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p = 0.2242, ANOVA — LS mean, SE of LS mean and p-value for treatment comparison are from ANOVA based on individual episodes with treatment as randomized, phase, and sequence as fixed factors and patient as random factor, using compound symmetry; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to .05], Standard Error of Mean 0.02

3. Secondary Outcome: Pain Intensity Difference (PID) at 10 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID10 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 10 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and 10 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | .35 (.05) | .29 (.05)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID10 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p = 0.0106, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [0.01 to .11], Standard Error of Mean 0.05

4. Secondary Outcome: Pain Intensity Difference (PID) at 30 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID30 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 30 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and 30 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | 2.10 (0.12) | 1.79 (0.12)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID30 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [.21 to .40], Standard Error of Mean 0.12

5. Secondary Outcome: Pain Intensity Difference (PID) at 45 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID45 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 45 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and 45 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | 3.13 (0.14) | 2.85 (0.14)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID45 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.18 to .37], Standard Error of Mean 0.14

6. Secondary Outcome: Pain Intensity Difference (PID) at 60 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID60 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 60 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and 60 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | 3.65 (0.15) | 3.48 (0.15)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID60 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p = 0.0002, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.08 to 0.27], Standard Error of Mean 0.15

7. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 5 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID5 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 5 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score.
Time Frame: Immediately pre-dose and 5 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 1.01 (4.50) | 0.73 (3.02)

8. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 10 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain. The PID10 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 10 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. This was assessed during the double-blind treatment period.
Time Frame: Immediately before treatment and 10 minutes after treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 4.83 (11.21) | 3.89 (8.30)

9. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 15 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed during the double-blind treatment period on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain. The PID15 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 15 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score.
Time Frame: Baseline (immediately pre-dose) and 15 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 12.38 (17.08) | 10.38 (15.43)

10. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 30 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID30 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 30 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score.
Time Frame: Pre-dose and 30 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 29.72 (21.30) | 25.03 (20.42)

11. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 45 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID45 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 45 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score.
Time Frame: Immediately pre-dose and 45 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 44.84 (23.36) | 40.49 (22.68)

12. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 60 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID60 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 60 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score.
Time Frame: Immediately pre-dose and 60 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 52.61 (24.33) | 49.47 (24.19)

13. Secondary Outcome: Sum of Pain Intensity Difference at 30 Minutes Post-treatment (SPID30)
Description: PI scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. SPID30 were derived from PID values. The SPID30 scores during the double-blind treatment phase were calculated as the time- weighted sum of the PID scores from 5 through 30 minutes,after the administration of study drug. SPID30 = (⅓ x PID5) + (⅓ x PID10) + (⅓ x PID15) + PID30. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: From 5 minutes after dosing through 30 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | 2.54 (0.17) | 2.16 (0.17)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [0.25 to 0.50]

14. Secondary Outcome: Sum of Pain Intensity Difference at 60 Minutes Post-treatment (SPID60)
Description: PI scores were assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine during the double-blind treatment period. The SPID60 was derived from PID values. The SPID60 scores during the double-blind treatment phase were calculated as the time- weighted sum of the PID scores from 5 through 60 minutes,after the administration of the study drug.
  SPID60 = SPID30 + PID45 + PID60. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: From 5 minutes after dosing through 60 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Units on a scale | 9.32 (0.44) | 8.50 (0.44)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [.55 to 1.10]

15. Secondary Outcome: Pain Relief (PR) Score at 5 Minutes Post-treatment
Description: The PR score 5 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 5 minutes after treatment
Population: Full Analysis Set defined as having at least one evaluable episode of breakthrough pain treated with FBT and at least one with oxycodone. An episode was evaluable if it had a valid pain intensity measurement immediately prior to drug administration. No imputation for missing breakthrough pain episodes, but LOCF was applied for missing PR scores.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Units on a scale | 0.11 (0.41) | 0.10 (0.36)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p = 0.5575, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

16. Secondary Outcome: Pain Relief Score at 10 Minutes Post-treatment
Description: The PR score 10 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 10 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Units on a scale | 0.32 (0.61) | 0.26 (0.49)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p = 0.0981, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

17. Secondary Outcome: Pain Relief Score at 15 Minutes Post-treatment
Description: The PR score 15 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 15 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Units on a scale | 0.68 (0.74) | 0.56 (0.70)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p = 0.0443, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

18. Secondary Outcome: Pain Relief Score at 30 Minutes Post-treatment
Description: The PR score 30 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 30 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Units on a scale | 1.48 (0.83) | 1.22 (0.81)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

19. Secondary Outcome: Pain Relief Score at 45 Minutes Post-treatment
Description: The PR score 45 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 45 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Units on a scale | 2.14 (0.82) | 1.90 (0.82)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

20. Secondary Outcome: Pain Relief Score at 60 Minutes Post-treatment
Description: The PR score 60 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 60 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Units on a scale | 2.44 (0.83) | 2.27 (0.82)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p = 0.0018, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

21. Secondary Outcome: Total Pain Relief at 60 Minutes (TOTPAR60)
Description: The mean TOTPAR at 60 minutes will be calculated for each episode as the weighted sum of Pain Relief (PR) scores (5-point Likert scale, 0 = none to 4 = complete) at each assessment of PR (during the double-blind treatment period) until 60 minutes after study drug administration, as follows:
  TOTPAR60 =(⅓ x PR5)+ (⅓ x PR10) +(⅓ x PR15)+ PR30 + PR45 + PR60. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: From 5 minutes to 60 minutes after dosing
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1335 | 1324
units on a scale | 6.43 (0.20) | 5.70 (0.20)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.74, 95% CI [0.58 to 0.90], Standard Error of Mean 0.20

22. Secondary Outcome: Percent Total Pain Relief at 60 Minutes Posttreatment (%TOTPAR)
Description: The PR score at set intervals after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete). The maximum TOTPAR score that could be achieved at 60 minutes is equal to 16; thus, %TOTPAR at 60 minutes is (TOTPAR60 /16) x 100.The % TOTPAR achieved 60 minutes after the administration of study drug was calculated during the double-blind treatment phase.
Time Frame: From 5 minutes through 60 minutes after study drug treatment
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Percentage change | 40.11 (16.32) | 35.59 (15.78)

23. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment - <= 5 Minutes
Description: Time to APR (subjective perception of any reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes which time to APR fell in that category was compared. Number of episodes where APR was achieved in 5 minutes or less was compared.
Time Frame: From time study drug was taken until 5 minutes after treatment
Population: Full Analysis Set defined by at least one episode of breakthrough pain treated with FBT and at least one with oxycodone. No imputation was done if subject never answered APR/MPR question. If responded only as no, remaining missing imputed as no. If at least 1 yes, remaining missing imputed as yes.
Measure: Number; unit: Episodes
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Episodes | 55 | 50
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Analysis is based on a generalized estimating equation model with treatment as a fixed effect and patient as a random effect. A logit link function and compound symmetry working correlation were applied in this model; Test type: Superiority or Other; p = 0.7012, Generalized Estimating Equation; Odds Ratio (OR) = 1.1464, 95% CI 2-sided [0.6 to 2.3]

24. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment <=10 Minutes
Description: Time to APR (subjective perception of any reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes which time to APR fell in that category was compared. Number of episodes where APR was achieved in 10 minutes or less was compared.
Time Frame: From study drug treatment until 10 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Episodes | 226 | 219
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.6545, Generalized Estimating Equation; Odds Ratio (OR) = 1.0704, 95% CI 2-sided [0.8 to 1.4]

25. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment <=15 Minutes
Description: Time to APR (subjective perception of any reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes which time to APR fell in that category was compared. Number of episodes where APR was achieved in 15 minutes or less was compared.
Time Frame: From study drug administration to 15 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Episodes | 515 | 451
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0407, Generalized Estimating Equation; Odds Ratio (OR) = 1.2544, 95% CI 2-sided [1.0 to 1.6]

26. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment <=30 Minutes
Description: Time to APR (subjective perception of any reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes which time to APR fell in that category was compared. Number of episodes where APR was achieved in 30 minutes or less was compared.
Time Frame: Time of study drug administration till 30 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: Breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (Breakthrough pain episodes) | 1342 | 1334
Episodes | 1004 | 877
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0007, Generalized Estimating Equation; Odds Ratio (OR) = 1.5745, 95% CI 2-sided [1.2 to 2.0]

27. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment <=45 Minutes
Description: Time to APR (subjective perception of any reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes which time to APR fell in that category was compared. Number of episodes where APR was achieved in 45 minutes or less was compared.
Time Frame: Time of study drug treatment until 45 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 1217 | 1150
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0372, Generalized Estimating Equation; Odds Ratio (OR) = 1.5828, 95% CI 2-sided [1.0 to 2.4]

28. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment <=60 Minutes
Description: Time to APR (subjective perception of any reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes which time to APR fell in that category was compared. Number of episodes where APR was achieved in 60 minutes or less was compared.
Time Frame: Time of study drug treatment until 60 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 1271 | 1239
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.3099, Generalized Estimating Equation; Odds Ratio (OR) = 1.3722, 95% CI 2-sided [0.7 to 2.5]

29. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment - <= 5 Minutes
Description: Time to MPR (subjective perception of meaningful reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point up to 60 minutes during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes which time to MPR fell in that category was compared.
Time Frame: From time study drug was taken until 5 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 21 | 26
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.5777, Generalized Estimating Equation; Odds Ratio (OR) = 0.8434, 95% CI 2-sided [.5 to 1.5]

30. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment <=10 Minutes
Description: Time to MPR(subjective perception of meaningful reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes which time to MPR fell in that category was compared. Number of episodes in which MPR was achieved in 10 minutes or less was compared.
Time Frame: Time of study drug treatment until 10 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 88 | 91
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.9567, Generalized Estimating Equation; Odds Ratio (OR) = 0.9860, 95% CI 2-sided [0.6 to 1.6]

31. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment <=15 Minutes
Description: Time to MPR(subjective perception of meaningful reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes which time to MPR fell in that category was compared. Number of episodes in which MPR was achieved in 15 minutes or less was compared.
Time Frame: Time of study drug administration until 15 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 230 | 212
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.4253, Generalized Estimating Equation; Odds Ratio (OR) = 1.1366, 95% CI 2-sided [0.8 to 1.6]

32. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment <=30 Minutes
Description: Time to MPR(subjective perception of meaningful reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes which time to MPR fell in that category was compared. Number of episodes in which MPR was achieved in 30 minutes or less was compared.
Time Frame: Time of study drug administration until 30 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 613 | 503
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0038, Generalized Estimating Equation; Odds Ratio (OR) = 1.4269, 95% CI 2-sided [1.1 to 1.8]

33. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment <=45 Minutes
Description: Time to MPR(subjective perception of meaningful reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes which time to MPR fell in that category was compared. Number of episodes in which MPR was achieved in 45 minutes or less was compared.
Time Frame: From study drug administration until 45 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 983 | 864
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0012, Generalized Estimating Equation; Odds Ratio (OR) = 1.5118, 95% CI [1.2 to 1.9]

34. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment <=60 Minutes
Description: Time to MPR(subjective perception of meaningful reduction in pain intensity) was measured by stopwatch and by scheduled questions at each time point during double-blind treatment period. No pain relief was defined as: patient indicated no pain relief experienced, rescue medication was used,or missing data. For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes which time to MPR fell in that category was compared. Number of episodes in which MPR was achieved in 60 minutes or less was compared.
Time Frame: Time of study drug administration until 60 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 1139 | 1047
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0074, Generalized Estimating Equation; Odds Ratio (OR) = 1.5826, 95% CI 2-sided [1.1 to 2.2]

35. Secondary Outcome: Use of Standard Rescue Medication
Description: Any use of standard rescue medication after the administration of study drug for relief of Breakthrough Pain (BTP) during the double-blind treatment phase was recorded in the patient's diary. The number of breakthrough pain episodes for which study drug treatment was administered and which required rescue medication use was recorded.
Time Frame: Throughout the double-blind treatment period
Population: as for outcome 15
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes | 39 | 41
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.8444, Generalized Estimating Equation; Odds Ratio (OR) = 1.0590, 95% CI 2-sided [0.6 to 1.9]

36. Secondary Outcome: Medication Performance Assessment 30 Minutes Post-treatment
Description: The medication performance assessment assessed study drug performance on a 5-point categorical scale of 0-4 (0=poor, 1=fair,2=good, 3=very good, 4=excellent) 30 minutes after administration of study drug during the double-blind treatment periods and for the first 5 BTP episodes after each visit during the open-label extension period were recorded in the patient's paper diary. Patients were asked "How well did your study medication perform in controlling this breakthrough pain episode?" The number of episodes rated for each category were recorded.
Time Frame: 30 minutes post-treatment
Population: as for outcome 15
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes
  Excellent | 49 | 16
  Very Good | 125 | 104
  Good | 378 | 304
  Fair | 416 | 391
  Poor | 341 | 489
  No Response | 33 | 30
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); Analysis is based on a generalized estimating equation model with treatment as a fixed effect and patient as a random effect. A cumulative logit link function and independent working correlation were applied in this model. Treatment differences for each time point were measured across all categories of responses; Test type: Superiority or Other; p < 0.0001, Generalized Estimating Equation; Odds Ratio (OR) = 1.6033, 95% CI 2-sided [1.4 to 1.8]

37. Secondary Outcome: Medication Performance Assessment 60 Minutes Post-treatment
Description: The medication performance assessment assessed study drug performance on a 5-point categorical scale of 0-4 (0=poor, 1=fair,2=good, 3=very good, 4=excellent) 60 minutes after administration of study drug during the double-blind treatment periods and for the first 5 BTP episodes after each visit during the open-label extension period were recorded in the patient's paper diary. Patients were asked "How well did your study medication perform in controlling this breakthrough pain episode?" The number of episodes rated for each category were recorded.
Time Frame: 60 minutes post-treatment
Population: as for outcome 15
Measure: Number; unit: Episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablet (FBT) | Immediate-release Oxycodone (OXY)
Number analyzed (Participants) | 137 | 137
Number analyzed (breakthrough pain episodes) | 1342 | 1334
Episodes
  Excellent | 160 | 119
  Very Good | 371 | 313
  Good | 508 | 565
  Fair | 181 | 179
  Poor | 92 | 136
  No Response | 30 | 22
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablet (FBT) vs Immediate-release Oxycodone (OXY); [analysis description as in outcome 36, analysis 1]; Test type: Superiority or Other; p < 0.0001, Generalized Estimating Equation; Odds Ratio (OR) = 1.3334, 95% CI 2-sided [1.2 to 1.5]

38. Secondary Outcome: Breakthrough Pain Preference Questionnaire
Description: The BTP preference questionnaire is a questionnaire used to measure patients' preference for FBT or immediate-release oxycodone for management of BTP. The question is used to determine a patient's preference between the study drugs given in the 2 double-blind treatment periods. The patient was asked to select 1 of the following: 1, a preference for study drug used in the 1st double-blind treatment period; 2, a preference for study drug used in the 2nd double-blind treatment period; or 3, no preference.
Time Frame: At Visit 6 ( up to 42 days depending upon how long it takes the patient to manage their BTP) after completion of both double-blind treatment periods.
Population: Double-blind safety analysis set: 143 subjects who received both study drugs in this crossover study completed the Breakthrough Pain Preference Questionnaire after completing treatment
Measure: Number; unit: Participants
Groups:
- Total: Includes all patients who participated in the double-blind treatment period and completed treatment.
  Immediate-release oxycodone or matching placebo at doses of 15, 30, 45, and 60 mg was self-administered by patients.
  During the 12-week open-label extension period, pts randomized to FBT treatment were initially dispensed single tablets at the dose found to be successful during the titration period.
Arm/Group | Total
Number analyzed (Participants) | 143
Participants
  Preferred FBT | 62
  Preferred Oxycodone | 46
  No Preference | 23
  Missing | 12

39. Secondary Outcome: Patient Global Impression of Change (PGIC) at Visit 7- 1 Month After Open Label Treatment
Description: The PGIC is a standardized self-report tool that measures the change in a patient's overall status rating since the start of the open-label extension period. The 7-point scale includes very much worse= -3, much worse= -2, minimally worse= -1, no change=0, minimally improved= +1, much improved= +2, and very much improved= +3. This was assessed 1 month after start of the open-label extension period.
Time Frame: One month after start of open-label treatment
Population: Open-Label Efficacy Assessment Set includes all subjects who were randomly assigned to the open-label treatments in the extension period and had an efficacy assessment for at least one of the efficacy questionnaires.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Groups:
- Fentanyl Buccal Tablet (FBT): FBT or matching placebo during the 2 double-blind treatment periods at doses of 200, 400, 600, and 800 mcg was self-administered by patients.
  Immediate-release oxycodone or matching placebo at doses of 15, 30, 45, and 60 mg was self-administered by patients.
  During the 12-week open-label extension period, pts randomized to FBT treatment were initially dispensed single tablets at the dose found to be successful during the titration period.
- Standard of Care (SOC): Randomized open-label extension to either FBT or alternate short-acting oral opioid therapy.
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 55 | 61
Unit on a scale | 1.5 (0.88) | 0.6 (0.99)

40. Secondary Outcome: Patient Global Impression of Change (PGIC) at Visit 8- 2 Months After Open Label Treatment
Description: The PGIC is a standardized self-report tool that measures the change in a patient's overall status rating since the start of the open-label extension period. The 7-point scale includes very much worse= -3, much worse= -2, minimally worse= -1, no change=0, minimally improved= +1, much improved= +2, and very much improved= +3. Here it was assessed 2 months after the start of the open-label extension period.
Time Frame: 2 months after start of open-label extension period
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 60
Units on scale | 1.5 (0.99) | 0.8 (0.99)

41. Secondary Outcome: Patient Global Impression of Change (PGIC) at Visit 9- 3 Months After Open Label Treatment
Description: The PGIC is a standardized self-report tool that measures the change in a patient's overall status rating since the start of the open-label extension period. The 7-point scale includes very much worse= -3, much worse= -2, minimally worse= -1, no change=0, minimally improved= +1, much improved= +2, and very much improved= +3. Here it was assessed 3 months after the start of the open-label extension period.
Time Frame: 3 months after start of open-label extension period
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 53 | 59
Units on scale | 1.7 (0.86) | 0.8 (1.09)

42. Secondary Outcome: Patient Global Impression of Change (PGIC) Endpoint
Description: The PGIC is a standardized self-report tool that measures the change in a patient's overall status rating since the start of the open-label extension period. The 7-point scale includes very much worse= -3, much worse= -2, minimally worse= -1, no change=0, minimally improved= +1, much improved= +2, and very much improved= +3. Here it was assessed at the conclusion of the open-label extension period.
Time Frame: At conclusion of open-label extension period
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 65 | 65
Units on a scale | 1.5 (1.02) | 0.9 (1.09)

43. Secondary Outcome: Clinician Global Impression of Change at Visit 7- 1 Month After Open Label Treatment
Description: The CGIC is a standardized tool that measures the change in a patient's overall status rating since the start of the open-label extension period, in the opinion of the clinician.
  The 7-point scale includes very much worse=-3, much worse=-2, minimally worse=-1,no change=0, minimally improved=+1, much improved=+2, and very much improved=+3. The CGIC was completed by the clinicians at visits 7, 8, and 9 (or early termination) which correspond to 1, 2, or 3 months after the start of the open-label extension period.
Time Frame: One month after start of open-label extension
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 57 | 63
Unit on a scale | 1.4 (0.79) | 0.6 (0.91)

44. Secondary Outcome: Clinician Global Impression of Change (CGIC) at Visit 8- 2 Months After Open Label Treatment
Description: The CGIC is a standardized tool that measures the change in a patient's overall status rating since the start of the open-label extension period, in the opinion of the clinician.
  The 7-point scale includes very much worse=-3, much worse=-2, minimally worse=-1,no change=0, minimally improved=+1, much improved=+2, and very much improved=+3. Here it was assessed 2 months after the start of the open-label extension period.
  The CGIC was completed by the clinicians at visits 7, 8, and 9 (or early termination).
Time Frame: Two months after start of open-label extension period
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 60
Units on a scale | 1.4 (0.96) | 0.7 (0.88)

45. Secondary Outcome: Clinician Global Impression of Change (CGIC) at Visit 9- 3 Months After Open Label Treatment
Description: The CGIC is a standardized tool that measures the change in a patient's overall status rating since the start of the open-label extension period, in the opinion of the clinician.
  The 7-point scale includes very much worse=-3, much worse=-2, minimally worse=-1,no change=0, minimally improved=+1, much improved=+2, and very much improved=+3. The CGIC was completed by the clinicians at visits 7, 8, and 9 (or early termination), which correspond to 1, 2, or 3 months after the start of the open-label extension period.
Time Frame: 3 months after start of open-label extension period
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 53 | 59
Units on a scale | 1.6 (0.81) | 0.7 (1.02)

46. Secondary Outcome: Clinician Global Impression of Change (CGIC)Endpoint
Description: The CGIC is a standardized tool that measures the change in a patient's overall status rating since the start of the open-label extension period, in the opinion of the clinician.
  The 7-point scale includes very much worse=-3, much worse=-2, minimally worse=-1,no change=0, minimally improved=+1, much improved=+2, and very much improved=+3. The CGIC was completed by the clinicians at visits 7, 8, and 9 (or early termination).
Time Frame: End of open-label extension period
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablet (FBT) | Standard of Care (SOC)
Number analyzed (Participants) | 65 | 65
Units on a scale | 1.4 (1.01) | 0.7 (1.05)

ADVERSE EVENTS:
Groups:
- Fentanyl Buccal Tablet: This was a crossover study in which subjects were first randomized to receive Fentanyl Buccal Tablet (FBT) or oxycodone in two titration periods of the study (titrated once with one drug and again with the other) and then were randomized to double-blind treatment first with one drug then the other. As a result, all subjects were exposed to both FBT and oxycodone at different times except for subjects who discontinued before the second titration period. 213 subjects began the first titration period and of those 17 discontinued before exposure to FBT. Including Titration Periods, Double-blind Treatment Periods and Open-Label Extension Periods 196 subjects had exposure to FBT
- Oxycodone: This was a crossover study in which subjects were first randomized to receive Fentanyl Buccal Tablet (FBT) or oxycodone in two titration periods of the study (titrated once with one drug and again with the other) and then were randomized to double-blind treatment first with one drug then the other. As a result, all subjects were exposed to both FBT and oxycodone at different times except for subjects who discontinued before the second titration period (they were only exposed to one drug). 213 subjects began the first titration period and of those 27 discontinued before exposure to oxycodone. Including Titration Periods, Double-blind Treatment Periods and Open-Label Extension Periods 186 subjects had exposure to oxycodone
- Standard of Care: 21 subjects received standard of care analgesics apart from oxycodone or FBT during the Open-Label Extension Period. Subjects who took oxycodone during SOC are listed under Oxycodone.
Arm/Group | Fentanyl Buccal Tablet | Oxycodone | Standard of Care
Serious Adverse Events (participants affected / at risk) | 4/196 | 3/186 | 1/21
Other Adverse Events (participants affected / at risk) | 45/196 | 42/186 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl Buccal Tablet (N=196) | Oxycodone (N=186) | Standard of Care (N=21)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Buccal Tablet (N=196) | Oxycodone (N=186) | Standard of Care (N=21)
Nausea (Gastrointestinal disorders) | 9 | 7 | 0
Vomiting (Gastrointestinal disorders) | 6 | 5 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 4 | 2
Influenza (Infections and infestations) | 3 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2
Liver function test abnormal (Investigations) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 2
Somnolence (Nervous system disorders) | 9 | 9 | 0
Headache (Nervous system disorders) | 8 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All unpublished information given to an investigator by Cephalon shall not be published or disclosed to a third party without the prior written consent of Cephalon.